CLINICAL TRIAL: NCT03386695
Title: Acceptability and Validity of Self Sampling for High Risk HPV Detection Among Women in Maharashtra
Acronym: HPV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Gauravi Ashish Mishra, Physician&Professor, Tata Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TMHPO 1686
Record Dates: First submitted 2017-04-18; First posted 2017-12-29 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer and HPV infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education by Pamphlets (Other): Half of the women in each group will be provided an information pamphlet on the risk factors, methods of early detection, prevention, signs and symptoms of cervical cancer and how to use the self samplers at home.
  Interventions: Other: Education by Pamphlets
- Health education programme (Other): Half of the women in each group will be invited to specially organised camps in their neighbourhood for Health Education and distribution of self samplers.
  Interventions: Other: Health education programme

INTERVENTIONS:
Other: Education by Pamphlets — Distribution of pamphlets with information of prevention and early detection of cervical cancer and written as well as pictorial depiction on how to collect cervical self sample for HPV detection.
  Arms: Education by Pamphlets
Other: Health education programme — Health education program explaining about prevention and early detection of cancer and education on method of collection of cervical self sample for HPV.
  Arms: Health education programme

SUMMARY:
The study goals are,

1. To determine the test characteristics (sensitivity, specificity, positive predictive value, negative predictive value, false positivity rates, false negativity rates) of health personnel collected and self collected HPV samples for Hybrid capture explained by two different methods (pamphlets/ health education programme).
2. To evaluate the agreement between self collected HPV samples and health personnel collected HPV samples for Hybrid capture with two different methods of education (pamphlets/ health education programme).
3. To study the attitudes, acceptability and barriers of self-collection of specimens for HPV DNA testing in three sub groups of population in Maharashtra with two different methods of education (pamphlets/ health education programme).
4. To determine the predictors of self-sampling preference.
5. To determine the Knowledge, Attitudes and Practices (KAP) regarding cervical cancer and HPV infection among these women in pre-intervention and post-intervention period.

DETAILED DESCRIPTION:
The three communities, urban slum area in Mumbai, urban non slum area in Mumbai and rural area in Raigad/ Thane district will be selected. The eligible women will be contacted by door to door visit and the purpose of the campaign will be explained to them. Informed consent will be obtained from those who are willing to participate in the study.

Step 1: They will be interviewed to collect the baseline Knowledge, Attitude and Practices (KAP) regarding cervical cancer, screening and HPV. The information will be recorded on a structured questionnaire.

Step 2: Half of the women in each group will be invited to specially organized camps in their neighborhood for Health Education and distribution of self samplers while the other half will be provided an information pamphlet on the risk factors, methods of early detection, prevention, signs and symptoms of cervical cancer and how to use the self samplers at home. Similar personal interviews, collection of used/unused self sampler and collection of HPV samples by health worker will be followed for both groups of women.

Intervention one: (Health Education Group) Detailed health education programme explaining them the risk factors, methods of early detection, prevention, signs and symptoms of cervical cancer will be conducted. They will be explained the importance of getting screened for cervical cancer and will be encouraged to undergo screening at any nearby screening centre. They will be given information regarding HPV self samplers and will be taught the method of its use and storage in detail. Any queries with this regard will be answered.

Intervention two: (Both Groups) HPV self samplers will be distributed free of cost to the women and the social workers will instruct them to return it to the clinic or will collect the samplers from their houses, either on the same day or the following day as per the convenience of the woman. For HPV self collection the participating women will be asked to collect the sample specimen as per instructions provided during the health education session/ pamphlets and store it at room temperature till the time of collection by the social worker. The willingness to use self sampler or refusal to use the HPV self sampler will be captured. Also, the reasons for their refusal shall be captured.

Step 3: (Both Groups) During the visit by social worker to collect the samples, the women will be again interviewed by the social worker for their experience about collecting the sample at home. Personal interviews will be conducted also to assess their acceptability of self sampling for HPV detection. Various queries regarding difficulties in obtaining, storing and transporting the samples as well as other potential factors likely to affect the acceptability of the self sampling methods will be assessed. Any injuries, barriers and motivators for self sampling will be recorded. The women who refuse to use self samplers at this stage will also be interviewed to understand the barriers. HPV sample will be collected by the health worker when the woman comes to return the sampler kit. It will also be collected for women who refuse self sampling but are ready for health worker collected sample.

Information about the post-intervention KAP regarding cervical cancer, screening and HPV will be again recorded on a structured questionnaire from all women.

Step 4: (Both Groups) HPV testing will be performed with the Hybrid Capture System II {Digene}, which detects 13 different high-risk HPV types {16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 68}. The test will run according to the manufacturer's protocol. HPV determination will be quantitative, and women with samples producing readings of one or more times the positive control (1pg/ml HPV DNA) will be considered as HPV test positive.

Step 5: (Both Groups) The reports of self sampling HPV will be distributed to the women after 15 days. The women who test positive on either test will be contacted personally by staff or by telephone and will be offered free Preventive Oncology check up, Colposcopy and necessary work up either at Tata Memorial Hospital. The women not willing to avail facility at TMH will be referred to the nearby municipal or private hospital offering these services.

The women who are positive or negative on colposcopy will undergo further diagnosis and management as per departmental service protocol. The health worker will co-ordinate between the field staff and the various departments at TMH. The health worker will submit the samples to the department of Microbiology at the TMH, will collect the reports and send it to the field social workers for distribution, will assist the HPV positive patients for further investigations and diagnosis at the TMH.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active women in the age group of 30-55 years in the selected areas.

Exclusion Criteria:

* Pregnant women
* Women having frank cervical cancer
* Women who have undergone total hysterectomy

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1600 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Agreement rate between health care personnel collected samples and self collected samples in these two groups. | 18 months
  Results obtained out of the health care personnel collected samples Vs self collected samples and correspondingly results of the test among women taught to use self samplers with the aid of pamphlets as compared to a well conducted health education programme will be evaluated using kappa statistics.

SECONDARY OUTCOMES:
Test characteristics of HPV self sample and health care worker collected sample by HPV HC 2. | 18 months
  sensitivity, specificity, positive predictive value, negative predictive value, false positive rate and false negative rate will be calculated for self collected HPV samples and health personnel collected HPV samples
Acceptability and barriers for self-collection of specimens for HPV DNA testing in an urban population. | 18 months
  The acceptability and barriers for self collection of specimens for HPV DNA test will be calculated by using multiple logistic regression analysis for various socio-demographic and risk factors and my recording of reasons for the same

CONTACTS AND LOCATIONS:
Overall Officials: Gauravi A Mishra, MD, Principal Investigator — Tata Memorial Hospital, Mumbai
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No